CLINICAL TRIAL: NCT04037592
Title: Dorsomedial Prefrontal Cortex and the Antidepressant Efficacy of Theta Burst Stimulation in Depressed Patients and Its Predictors
Brief Title: Dorsomedial Prefrontal Cortex and the Antidepressant Efficacy of Theta Burst Stimulation in Depressed Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2018-07-011C
Record Dates: First submitted 2019-07-26; First posted 2019-07-30 (Actual); Last update posted 2022-08-31 (Actual); Status verified 2022-08

CONDITIONS: Treatment Resistant Depression
MeSH Terms: conditions — Depressive Disorder, Treatment-Resistant

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Active standardized iTBS-DMPFC (Experimental): This active group will receive standardized dosage of intermittent theta-burst on dorsomedial prefrontal cortex(DMPFC)
  Interventions: Device: Active standardized iTBS-DMPFC
- Active high-dosage iTBS-DMPFC (Experimental): This active group will receive high dosage of intermittent theta-burst on dorsomedial prefrontal cortex(DMPFC)
  Interventions: Device: Active high-dosage iTBS-DMPFC
- Sham standardized iTBS-DMPFC or high-dosage iTBS-DMPFC (Sham Comparator): Patients in the sham group will receive the same standardized or high-dosage iTBS performing by a sham coil
  Interventions: Device: Sham standardized iTBS-DMPFC or high-dosage iTBS-DMPFC

INTERVENTIONS:
Device: Active standardized iTBS-DMPFC — Participants in the standardized dosage(600 pulse) of intermittent TBS(iTBS) active stimulation group will receive 3-week three-pulse 50-Hz bursts administered every 200 milliseconds (at 5 Hz) at an intensity of 80% active motor threshold (MT) to bilateral DMPF, twice a day. Bilateral side DMPFC will be targeted by MRI-neuronavigation system. Stimulation will be delivered to the DMPFC using a Magstim stimulator.
  Arms: Active standardized iTBS-DMPFC
Device: Active high-dosage iTBS-DMPFC — Participants in the standardized dosage(1800pulse) of intermittent TBS(iTBS) active stimulation group will receive 3-week three-pulse 50-Hz bursts administered every 200 milliseconds (at 5 Hz) at an intensity of 80% active motor threshold (MT) to bilateral DMPF, twice a day. Bilateral side DMPFC will be targeted by MRI-neuronavigation system. Stimulation will be delivered to the DMPFC using a Magstim stimulator.
  Arms: Active high-dosage iTBS-DMPFC
Device: Sham standardized iTBS-DMPFC or high-dosage iTBS-DMPFC — Half of the patients in the sham group received 3-week the same standardized iTBS parameter stimulation (standardized sham-iTBS), and the other half received the same high dosage iTBS parameter stimulation using a sham coil (high dosage sham-rTMS), which also improved the blinding process
  Arms: Sham standardized iTBS-DMPFC or high-dosage iTBS-DMPFC

SUMMARY:
This study evaluates an association between different dosage and the antidepressant efficacy of theta burst stimulation in patients with treatment-resistant depression. In a double-blind design, All patients are randomized to three groups, i.e. standardized dosage intermittent theta-burst stimulation treatment, high dosage intermittent theta-burst stimulation treatment or sham treatment.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, 21 to 70 years of age.
* Diagnosed with the recurrent Major depressive disorder (MDD) and currently having a Major Depressive Episode (MDE)
* Participants failed to respond to at least one adequate antidepressant treatment in their current episode
* Participants have a Clinical Global Impression - Severity score of at least 4 and a total score of at least 18 on the Hamilton Depression Rating Scale (HDRS-17) at both screening and baseline visits ( Day -14 and Day 0)
* Participants must discontinue their antidepressant medications at least for one week ( at least two weeks if Fluoxetine) prior to the TMS intervention and keep antidepressant-free during the study duration.
* Participants also failed to respond to one complete left-sided DLPFC 10Hz rTMS/piTBS treatment course.

Exclusion Criteria:

* a lifetime psychiatric history of bipolar disorder, schizophrenia, psychotic disorders, or organic mental disorder including substance abuse and dependence (based on DSM-IV criteria)
* Participants with a lifetime medical history of major systemic illness and clinically significantly abnormal screening examination that might affect safety, study participation, or confound interpretation of study results.
* Participants with a lifetime medical history of neurological disorder records (e.g., stroke, seizure, traumatic brain injury, post brain surgery), brain implants (neurostimulators), cardiac pacemakers
* Women with breastfeeding or pregnancy
* Participants with a current strong suicidal risk (i.e., a score of 4 on item 3 of the HDRS-17)

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2019-07-24 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2021-01-31 (Actual)

PRIMARY OUTCOMES:
Percentage change in 17-item Hamilton Depression Rating Scale | Baseline, Week 1, Week 2, Week 3, Week 15(three-month after brain stimulation), Week 27(Six-month after brain stimulation)
  the altered percentage of 17-item Hamilton Depression Rating Scale (range, 0 to 52, with higher scores indicating more depression)

SECONDARY OUTCOMES:
Response rate after 3-week treatment at the end of iTBS sessions and three and six month after. | Baseline, Week 1, Week 2, Week 3, Week 15(three-month after brain stimulation), Week 27(Six-month after brain stimulation)
  improvement > 50 % of 17-item Hamilton Depression Rating Scale (range, 0 to 52, with higher scores indicating more depression)
Remission rate after 3-week treatment | Baseline, Week 1, Week 2, Week 3, Week 15(three-month after brain stimulation), Week 27(Six-month after brain stimulation)
  17-item Hamilton Depression Rating Scale ≤7 (range, 0 to 52, with higher scores indicating more depression)
Changes in Clinical Global Index | Baseline, Week 1, Week 2, Week 3
  Clinical Global Index
Changes in depression severity, rated by self-reported | Baseline, Week 1, Week 2, Week 3
  Depression and Somatic Symptoms Scale, range from 0 to 66 with higher scores indicating more depressive and somatic symptom.
Changes in Young Mania Rating Scale | Baseline, Week 1, Week 2, Week 3
  Young Mania Rating Scale, range from 0 to 60 with higher scores indicating more severe manic symptoms.
Baseline treatment refractory level and the further antidepressant efficacy of brain stimulation | Baseline, Week 3
  Maudsley staging method
Baseline brain connectivity and the further antidepressant efficacy of brain stimulation | Baseline, Week 3
  baseline functional MRI
the change of brain connectivity after 3-week iTBS treatment | Baseline, Week 3
  the change in brain connectivity
Baseline Life event stress scale and the further antidepressant efficacy of brain stimulation | Baseline, Week 3
  Life event stress scale,range from 0 to 1467 with higher scores indicating more life event stress.
Changes in EEG band before and after brain stimulation | Day 1(pre-RECT, post RECT, post 1st treatment, pre-30th treatment)
  Perform rostral anterior cingulate cortex(rACC)-engaging cognitive task(RECT) before 1-st treatment
Baseline single-pulse stimulation and the further antidepressant efficacy of brain stimulation | Baseline, Week 3
  baseline single-pulse stimulation
Changes in single-pulse stimulation before and after brain stimulation | Baseline, Week 3
  the change in single-pulse stimulation
Baseline paired-pulse stimulation and the further antidepressant efficacy of brain stimulation | Baseline, Week 3
  baseline paired-pulse stimulation
Changes in paired-pulse stimulation before and after brain stimulation | Baseline, Week 3
  the change in paired-pulse stimulation
Change in anxiosomatic cluster symptoms derived 17-item Hamilton Depression Rating Scale | Baseline, Week 1, Week 2, Week 3
  the altered anxiosomatic cluster symptoms (range, 0 to 26, with higher scores indicating more severe anxiosomatic symptoms).The anxiosomatic cluster symptoms comprised nine items derived from HDRS-17: early insomnia, middle insomnia, slowness or retardation, psychic anxiety, autonomic anxiety, gastrointestinal symptoms, somatic symptoms, genital symptoms, and hypochondriasis.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Psychiatry, Taipei Veterans General Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cheng CM, Li CT, Jeng JS, Chang WH, Lin WC, Chen MH, Bai YM, Tsai SJ, Su TP. Antidepressant effects of prolonged intermittent theta-burst stimulation monotherapy at the bilateral dorsomedial prefrontal cortex for medication and standard transcranial magnetic stimulation-resistant major depression: a three arm, randomized, double blind, sham-controlled pilot study. Eur Arch Psychiatry Clin Neurosci. 2023 Oct;273(7):1433-1442. doi: 10.1007/s00406-022-01523-4. Epub 2022 Dec 9. PMID 36484844